CLINICAL TRIAL: NCT05859516
Title: Application of Point-of-care Ultrasound in Rapid Assessment of Cardiac Arrest Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022003
Record Dates: First submitted 2023-03-24; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2022-09

CONDITIONS: Cardiac Arrest; Point-of-care Ultrasound; Cardiopulmonary Resuscitation
Keywords: Cardiac Arrest; Point-of-care Ultrasound; cardiopulmonary resuscitation quality
MeSH Terms: conditions — Heart Arrest | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — whole blood; serum; urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Ultrasound
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Every time checking pulse, evaluate the carotid artery compressibility and blood flow of peripheral arteries by ultrasound，compared with EtCO2.

SUMMARY:
To quickly assess the patient's cardiac function and structure through ultrasound

DETAILED DESCRIPTION:
Monitor the peripheral arterial pulse and flow velocity, monitor the patient's lung and diaphragm muscle movement, monitor the patient's optic nerve sheath and cerebral blood flow, observe the morphology and blood flow of the liver and kidney and other parenchymal organs, Comprehensive evaluation of patient resuscitation quality.

For patients with cardiac arrest undergoing Cardio Pulmonary Resuscitation (CPR), the above monitoring was completed by ultrasound, and compared with the parameters obtained by end-expiratory carbon dioxide (ETCO2) and compression feedback device, to evaluate the feasibility of ultrasound to evaluate the quality of CPR. After the reliability evaluation was completed, parameters were further used to guide CPR quality improvement through ultrasound, end-expiratory carbon dioxide (ETCO2), and compression feedback device.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate and sign a written informed consent;
* Male or female above 18;
* Patients who are sent to the emergency room of our hospital with symptoms of "cardiopulmonary resuscitation";

Exclusion Criteria:

* There is trauma in the ultrasound examination site and it is not suitable for ultrasound examination;
* Entering the emergency room without vital signs for more than 30 minutes;
* The appearance of corpse corpses;
* There is life-threatening and irreversible damage;
* Other investigators consider it inappropriate and the patient or family member refuses;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The correlation between return of spontaneous circulation rate and peripheral blood flow through study completion, an average of 1 hour. | through study completion, an average of 1 hour.
  For patients with cardiac arrest undergoing CPR, Peripheral arterial blood flow monitoring was completed by ultrasound, and compared with treturn of spontaneous circulation rate .
  Bilateral carotid blood flow velocity:
  1. Peak systolic velocity, PSV, cm/s
  2. End diastolic velocity, EDV,cm/s
  3. Resistance index, RI
  4. Pulsatility index, PI Bilateral femoral artery blood flow velocity
  1) Peak systolic velocity, PSV, cm/s 2) End diastolic velocity, EDV,cm/s 3) Resistance index, RI 4) Pulsatility index, P

CONTACTS AND LOCATIONS:
Overall Officials: Jian Xia, Dr., Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandor A, Fuller G, Essat M, Sabir L, Holt C, Buckley Woods H, Chatha H. Individual risk factors predictive of major trauma in pre-hospital injured older patients: a systematic review. Br Paramed J. 2022 Mar 1;6(4):26-40. doi: 10.29045/14784726.2022.03.6.4.26. PMID 35340581
- [Background] Mederos MA, Reber HA, Girgis MD. Acute Pancreatitis: A Review. JAMA. 2021 Jan 26;325(4):382-390. doi: 10.1001/jama.2020.20317. PMID 33496779
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Reynolds JC, Nicholson T, O'Neil B, Drennan IR, Issa M, Welsford M; Advanced Life Support Task Force at the International Liaison Committee on Resuscitation ILCOR. Diagnostic test accuracy of point-of-care ultrasound during cardiopulmonary resuscitation to indicate the etiology of cardiac arrest: A systematic review. Resuscitation. 2022 Mar;172:54-63. doi: 10.1016/j.resuscitation.2022.01.006. Epub 2022 Jan 19. PMID 35065210
- [Background] Montoya J, Stawicki SP, Evans DC, Bahner DP, Sparks S, Sharpe RP, Cipolla J. From FAST to E-FAST: an overview of the evolution of ultrasound-based traumatic injury assessment. Eur J Trauma Emerg Surg. 2016 Apr;42(2):119-26. doi: 10.1007/s00068-015-0512-1. Epub 2015 Mar 14. PMID 26038031
- [Background] Keikha M, Salehi-Marzijarani M, Soldoozi Nejat R, Sheikh Motahar Vahedi H, Mirrezaie SM. Diagnostic Accuracy of Rapid Ultrasound in Shock (RUSH) Exam; A Systematic Review and Meta-analysis. Bull Emerg Trauma. 2018 Oct;6(4):271-278. doi: 10.29252/beat-060402. PMID 30402514
- [Background] Dicker SA. Lung Ultrasound for Pulmonary Contusions. Vet Clin North Am Small Anim Pract. 2021 Nov;51(6):1141-1151. doi: 10.1016/j.cvsm.2021.07.001. Epub 2021 Sep 11. PMID 34521570
- [Background] Lichtenstein D. Fluid administration limited by lung sonography: the place of lung ultrasound in assessment of acute circulatory failure (the FALLS-protocol). Expert Rev Respir Med. 2012 Apr;6(2):155-62. doi: 10.1586/ers.12.13. PMID 22455488
- [Background] Kang SY, Jo IJ, Lee G, Park JE, Kim T, Lee SU, Hwang SY, Shin TG, Kim K, Shim JS, Yoon H. Point-of-care ultrasound compression of the carotid artery for pulse determination in cardiopulmonary resuscitation. Resuscitation. 2022 Oct;179:206-213. doi: 10.1016/j.resuscitation.2022.06.025. Epub 2022 Jul 2. PMID 35792305
- [Background] Sheak KR, Wiebe DJ, Leary M, Babaeizadeh S, Yuen TC, Zive D, Owens PC, Edelson DP, Daya MR, Idris AH, Abella BS. Quantitative relationship between end-tidal carbon dioxide and CPR quality during both in-hospital and out-of-hospital cardiac arrest. Resuscitation. 2015 Apr;89:149-54. doi: 10.1016/j.resuscitation.2015.01.026. Epub 2015 Jan 30. PMID 25643651
- [Background] Genbrugge C, Dens J, Meex I, Boer W, Eertmans W, Sabbe M, Jans F, De Deyne C. Regional Cerebral Oximetry During Cardiopulmonary Resuscitation: Useful or Useless? J Emerg Med. 2016 Jan;50(1):198-207. doi: 10.1016/j.jemermed.2015.03.043. Epub 2015 Sep 26. PMID 26412107
- [Background] Reynolds JC, Issa MS, C Nicholson T, Drennan IR, Berg KM, O'Neil BJ, Welsford M; Advanced Life Support Task Force of the International Liaison Committee on Resuscitation. Prognostication with point-of-care echocardiography during cardiac arrest: A systematic review. Resuscitation. 2020 Jul;152:56-68. doi: 10.1016/j.resuscitation.2020.05.004. Epub 2020 May 11. PMID 32437781
- [Background] Kedan I, Ciozda W, Palatinus JA, Palatinus HN, Kimchi A. Prognostic value of point-of-care ultrasound during cardiac arrest: a systematic review. Cardiovasc Ultrasound. 2020 Jan 13;18(1):1. doi: 10.1186/s12947-020-0185-8. PMID 31931808